CLINICAL TRIAL: NCT06658886
Title: Comparison of the Efficacy of Ultrasound-Guided Corticosteroid Injection and Paraffin Therapy in Carpal Tunnel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH9
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paraffin treatment group: Patients with carpal tunnel syndrome who have received paraffin therapy
  Interventions: Other: No intervention
- Injection group: Patients with carpal tunnel syndrome who have applied ultrasound-guided steroid injection
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to compare the efficacy of paraffin therapy, a physical therapy modality, and ultrasound-guided corticosteroid injection in the treatment of carpal tunnel syndrome, the most common entrapment neuropathy. By doing so, the study will evaluate the effectiveness and feasibility of these two alternative, low-side-effect treatments for managing this frequently encountered condition.

DETAILED DESCRIPTION:
A total of 46 patients, aged 18-65, diagnosed with mild to moderate carpal tunnel syndrome based on electrophysiological studies, will be included in the study.Pain levels will be assessed using the Visual Analog Scale (VAS), and functional impairment will be measured with the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ). Electrophysiological evaluations will be performed by a neurology specialist at the 1st and 3rd month follow-ups outside of working hours and without being billed to the Social Security Institution (SGK). VAS, BCTQ scores, and electrophysiological parameters will be evaluated at baseline, and at the 4th and 12th-week follow-ups post-treatment. Electrophysiological measurements will include median nerve distal motor latency (MMNDL), median nerve distal sensory latency (MNSDL), sensory nerve conduction velocity (SNCV), compound muscle action potential (CMAP), and sensory nerve action potential (SNAP) amplitudes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65.
* Diagnosed with mild to moderate carpal tunnel syndrome based on electrophysiological studies.
* Received either ultrasound-guided corticosteroid injection or paraffin therapy.
* Symptoms persisting for at least 3 months.

Exclusion Criteria:

* Diagnosis of other conditions causing neuropathic symptoms (e.g., polyneuropathy, brachial plexopathy, thoracic outlet syndrome).
* History of previous injection or surgery for carpal tunnel syndrome.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mild and moderate carpal tunnel syndrome
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS): | 0 day, 4th week and 12th week
  The VAS will be used to measure pain intensity. Patients will mark their pain level on a 10 cm scale, where 0 represents "no pain" and 10 represents the "worst imaginable pain." This will be evaluated at baseline, and at the 4th and 12th weeks post-treatment.
Boston Carpal Tunnel Syndrome Questionnaire Symptom Severity Scale (BCTQ-SSS) | 0 day, 4th week and 12th week
  The SSS assesses the severity of carpal tunnel symptoms such as pain, tingling, and numbness. The total score for this scale ranges from a minimum of 11 to a maximum of 55. A lower score indicates mild or no symptoms, while a higher score suggests more severe symptoms. As the score increases, the severity of symptoms worsens, with a score closer to 55 reflecting a significantly greater impact on daily life.
Boston Carpal Tunnel Syndrome Questionnaire Functional Status Scale (BCTQ-FSS) | 0 day, 4th week and 12th week
  The SSS assesses the severity of carpal tunnel symptoms such as pain, tingling, and numbness. The total score for this scale ranges from a minimum of 11 to a maximum of 55. A lower score indicates mild or no symptoms, while a higher score suggests more severe symptoms. As the score increases, the severity of symptoms worsens, with a score closer to 55 reflecting a significantly greater impact on daily life.

SECONDARY OUTCOMES:
Median nerve distal motor latency | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Median nerve distal sensory latency | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Sensory nerve conduction velocity | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Motor nerve conduction velocity | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Sensory nerve action potential amplitude | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation
Motor nerve action potential amplitude | 0 day, 4th week and 12th week
  It is a finding from electrophysiological evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No